CLINICAL TRIAL: NCT01009060
Title: A Randomised Double-blind, Placebo Controlled, Parallel Group Study to Evaluate the Cognitive Enhancing Effect of GSK239512 in Stable Patients With Schizophrenia
Brief Title: Study to Evaluate the Efficacy and Safety of GSK239512 in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113147
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
Keywords: H3 Antagonist; Schizophrenia; double blind; Histamine; randomised; placebo controlled; Cognition
MeSH Terms: conditions — Schizophrenia | interventions — GSK239512

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK239512 (Experimental): Repeat dose.
  Interventions: Drug: GSK239512
- Placebo (Placebo Comparator): Repeat dose. Placebo to match GSK239512
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK239512 — Histamine H3 Antagonist
  Arms: GSK239512
Drug: Placebo — Placebo to match GSK239512
  Arms: Placebo

SUMMARY:
This study aims to evaluate the cognitive enhancing effects and tolerability of GSK239512 compared to placebo in patients with schizophrenia

DETAILED DESCRIPTION:
This is a 7-week, Phase II, multi-centre, randomised, double-blind, placebo-controlled, parallel group design study in male and female subjects with schizophrenia who are stabilised on antipsychotic medication. Subjects will be randomised to receive either GSK239512 or placebo for 7 weeks. They will undergo weekly review of safety, tolerability and cognitive performance measures.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Schizophrenia
2. No acute exacerbation of symptoms requiring hospital admission or step up care in the previous six months.
3. Not on any symptomatic treatment for cognition

Exclusion Criteria:

1. Poses a significant homicidal or suicidal risk or evidence of previous homicidal or suicidal risk.
2. Co-morbid psychiatric or significant physical illness
3. Alcohol or drug abuse or dependence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2011-08-10 (Actual); Study Completion 2011-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (14):
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Catonsville, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Jamaica Plain, Massachusetts
  - GSK Investigational Site, Mount Laurel, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Butner, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Jarskog LF, Lowy MT, Grove RA, Keefe RS, Horrigan JP, Ball MP, Breier A, Buchanan RW, Carter CS, Csernansky JG, Goff DC, Green MF, Kantrowitz JT, Keshavan MS, Laurelle M, Lieberman JA, Marder SR, Maruff P, McMahon RP, Seidman LJ, Peykamian MA. A Phase II study of a histamine H(3) receptor antagonist GSK239512 for cognitive impairment in stable schizophrenia subjects on antipsychotic therapy. Schizophr Res. 2015 May;164(1-3):136-42. doi: 10.1016/j.schres.2015.01.041. Epub 2015 Feb 24. PMID 25728831
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 centers in the United States from 1 December 2009 to 10 August 2011. Study included d-amphetamine therapeutic challenge (dropped in amendment 2), treatment period of 7 weeks (4 weeks titration and 3 weeks of maintenance) and follow up visit approximately 7-10 days following their last dose of study medication.
Pre-assignment Details: A total of 118 participants (par.) were screened. Out of these 50 participants were randomized. Out of these, safety population consisted of 50 participants and intent-to-treat (ITT) population consisted of 46 participants.
Groups:
- Placebo: Par. received oral placebo tablet matching with GSK239512 once daily for a period of 7 weeks.
- GSK239512: Par. received oral GSK239512 once daily for a period of 7 weeks (4 weeks titration and 3 weeks at maintenance). Par. started at a daily dose of 10 micrograms (μg) GSK239512 and titrated up weekly through successive dose levels of 20 μg, 40 μg up to a maximum dose of 80 μg according to the titration regimen.
Period: Overall Study
Arm/Group | Placebo | GSK239512
Started | 25 | 25
Completed | 21 | 20
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristic data is presented for ITT population which consisted of all participants randomized to treatment, who had taken at least one dose of investigational product and who had at least one post-Baseline CogState Schizophrenia Battery (CSSB) assessment during the on-treatment phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK239512 | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.1 (9.54) | 38.2 (13.10) | 39.2 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 19 | 17 | 36
Race/Ethnicity, Customized [Number; unit: Number]
  African American/African Heritage | 11 | 11 | 22
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 13 | 8 | 21
  Mixed Race | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Composite Score of CSSB Following Dosing With GSK239512
Description: The CSSB is a computerized battery with following domains (score range): Verbal memory (0-75), working memory (0-28), motor speed (0-100), verbal fluency, attention and speed of information processing (0-110) and executive functions with higher score representing better performance. Two Baseline CSSB testing were conducted; the first on the day prior to commencing dosing (Day -1) and the other test pre-dose on Day 1: the average of the two tests was used as Baseline. Change from Baseline was calculated as score at a given time minus score at Baseline. For each individual task from the CSSB, the Baseline was calculated as the mean of the second screening assessment and the Day 1 pre-dose assessment. A composite score was calculated by averaging all the measures, and then calculating a z-score of the composite. Higher the composite score, better is the performance. Z-score is the measure of standard deviation away from the mean score.
Time Frame: Baseline and up to Week 7
Population: ITT Population. Only those participants available at the specified time points were analyzed. Par. recruited under protocol amendment 2 were not assessed at Weeks 1, 3, 5 or 6 and hence the number of par. at these visits are lower.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 24 | 22
Scores on a scale
  Week 1: number analyzed (Participants) | 12 | 10
  Week 1 | 0.065 (0.0606) | 0.016 (0.1342)
  Week 2: number analyzed (Participants) | 23 | 21
  Week 2 | 0.086 (0.0814) | 0.104 (0.0682)
  Week 3: number analyzed (Participants) | 12 | 9
  Week 3 | 0.076 (0.0816) | -0.012 (0.1139)
  Week 4: number analyzed (Participants) | 22 | 20
  Week 4 | 0.157 (0.0859) | 0.068 (0.0901)
  Week 5: number analyzed (Participants) | 12 | 9
  Week 5 | 0.099 (0.0675) | 0.184 (0.1057)
  Week 6: number analyzed (Participants) | 12 | 9
  Week 6 | -0.001 (0.1234) | 0.194 (0.1539)
  Week 7: number analyzed (Participants) | 22 | 19
  Week 7 | 0.004 (0.1106) | 0.107 (0.1105)
Statistical Analysis 1: Comparison: Placebo vs GSK239512; Week 1; Test type: Superiority or Other; p = 0.7239, Mixed Model Repeated Measure; Mean Difference (Net) = -0.049, 90% CI 2-sided [-0.288 to 0.190]
Statistical Analysis 2: Comparison: Placebo vs GSK239512; Week 2; Test type: Superiority or Other; p = 0.8351, Mixed Model Repeated Measure; Mean Difference (Net) = 0.018, 90% CI 2-sided [-0.127 to 0.163]
Statistical Analysis 3: Comparison: Placebo vs GSK239512; Week 3; Test type: Superiority or Other; p = 0.4541, Mixed Model Repeated Measure; Mean Difference (Net) = -0.088, 90% CI 2-sided [-0.287 to 0.110]
Statistical Analysis 4: Comparison: Placebo vs GSK239512; Week 4; Test type: Superiority or Other; p = 0.4148, Mixed Model Repeated Measure; Mean Difference (Net) = -0.089, 90% CI 2-sided [-0.272 to 0.093]
Statistical Analysis 5: Comparison: Placebo vs GSK239512; Week 5; Test type: Superiority or Other; p = 0.3887, Mixed Model Repeated Measure; Mean Difference (Net) = 0.086, 90% CI 2-sided [-0.082 to 0.254]
Statistical Analysis 6: Comparison: Placebo vs GSK239512; Week 6; Test type: Superiority or Other; p = 0.2594, Mixed Model Repeated Measure; Mean Difference (Net) = 0.195, 90% CI 2-sided [-0.093 to 0.484]
Statistical Analysis 7: Comparison: Placebo vs GSK239512; Week 7; Test type: Superiority or Other; p = 0.4778, Mixed Model Repeated Measure; Mean Difference (Net) = 0.103, 90% CI 2-sided [-0.139 to 0.344]

2. Secondary Outcome: Change From Baseline in Composite Score of Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) at Week 7
Description: MCCB measures functioning across various cognitive domains and is comprised of ten tests that assess seven cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition). Its measurements are based on timed paper-and-pencil, computerized, and orally-administered tests, as well as spatial tests using geometric cubes. MCCB composite T scores are between 40 and 60 (normal range) and < 40 (below normal range). Higher scores indicate better performance. The Baseline was calculated as the mean of the second screening assessment and the Day 1 pre-dose assessment. If either measurement meant to be used in the mean was missing, then the Baseline value was the non-missing assessment. If both were missing, then Baseline was considered missing and the task was excluded from the analysis. Change from Baseline was calculated as score at a given time post Baseline minus score at Baseline.
Time Frame: Baseline and Week 7
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 22 | 19
Scores on a scale | 1.108 (1.8759) | 0.371 (1.7801)
Statistical Analysis 1: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.6947, ANCOVA; Mean Difference (Net) = -0.737, 90% CI 2-sided [-3.884 to 2.409]

3. Secondary Outcome: Change From Baseline in Individual Cognitive Domain Scores in CSSB at Week 7
Description: as for outcome 1
Time Frame: Baseline and Week 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 24 | 22
Scores on a scale
  Speed of Processing/Simple Reaction Time: number analyzed (Participants) | 22 | 18
  Speed of Processing/Simple Reaction Time | 0.541 (0.1628) | 0.289 (0.1391)
  Attention/Vigilance: number analyzed (Participants) | 22 | 18
  Attention/Vigilance | 0.067 (0.1756) | 0.246 (0.1932)
  Working Memory: number analyzed (Participants) | 22 | 17
  Working Memory | 0.021 (0.2030) | 0.412 (0.2164)
  Visual Learning: number analyzed (Participants) | 22 | 19
  Visual Learning | -0.198 (0.2414) | 0.081 (0.1699)
  Verbal Learning: number analyzed (Participants) | 22 | 19
  Verbal Learning | -0.558 (0.2853) | -0.160 (0.2339)
  Reasoning/Problem Solving: number analyzed (Participants) | 22 | 19
  Reasoning/Problem Solving | 0.016 (0.1168) | 0.192 (0.1085)
  Social Cognition: number analyzed (Participants) | 20 | 19
  Social Cognition | -0.431 (0.1544) | -0.401 (0.1339)
  Working Memory (Two-Back Memory): number analyzed (Participants) | 22 | 17
  Working Memory (Two-Back Memory) | 0.247 (0.1862) | 0.316 (0.2374)
Statistical Analysis 1: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.1399, Mixed Model Repeated Measure; Mean Difference (Net) = -0.252, 90% CI 2-sided [-0.535 to 0.030] — For Speed of Processing/Simple Reaction Time
Statistical Analysis 2: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.3992, Mixed Model Repeated Measure; Mean Difference (Net) = 0.179, 90% CI 2-sided [-0.176 to 0.534] — For Attention/Vigilance
Statistical Analysis 3: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.1547, Mixed Model Repeated Measure; Mean Difference (Net) = 0.391, 90% CI 2-sided [-0.063 to 0.845] — For Working Memory
Statistical Analysis 4: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.2531, Mixed Model Repeated Measure; Mean Difference (Net) = 0.279, 90% CI 2-sided [-0.127 to 0.685] — For Visual Learning
Statistical Analysis 5: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.2417, Mixed Model Repeated Measure; Mean Difference (Net) = 0.398, 90% CI 2-sided [-0.167 to 0.963] — For Verbal Learning
Statistical Analysis 6: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.2069, Mixed Model Repeated Measure; Mean Difference (Net) = 0.177, 90% CI 2-sided [-0.055 to 0.409] — For Reasoning/Problem Solving
Statistical Analysis 7: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.8645, Mixed Model Repeated Measure; Mean Difference (Net) = 0.030, 90% CI 2-sided [-0.262 to 0.322] — For Social Cognition
Statistical Analysis 8: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.7873, Mixed Model Repeated Measure; Mean Difference (Net) = 0.069, 90% CI 2-sided [-0.364 to 0.503] — For Working Memory (Two-Back Memory)

4. Secondary Outcome: Change From Baseline in Individual Cognitive Domain Scores in MCCB at Week 7
Description: MCCB measures functioning across various cognitive domains and is comprised of ten tests that assess seven cognitive domains (speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition) Its measurements are based on timed paper-and-pencil, computerized, and orally-administered tests, as well as spatial tests using geometric cubes. MCCB composite T scores are between 40 and 60 (normal range) and < 40 (below normal range). Higher scores indicate better performance. The Baseline was calculated as the mean of the second screening assessment and the Day 1 pre-dose assessment. If either measurement meant to be used in the mean was missing, then the Baseline value was the non-missing assessment. If both were missing, then Baseline was considered missing and the task was excluded from the analysis. Change from Baseline was calculated as score at a given time post Baseline minus score at Baseline.
Time Frame: Baseline and Week 7
Population: ITT Population. Only those participants at indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 22 | 19
T-scores
  Speed of Processing | 2.045 (1.7359) | -1.979 (1.6030)
  Attention/Vigilance | -0.111 (2.3028) | -2.351 (2.1303)
  Working Memory | 3.368 (2.0677) | 1.330 (1.9086)
  Visual Learning | -0.718 (2.3868) | -1.464 (2.2060)
  Verbal Learning | -1.174 (2.1772) | 1.938 (2.1123)
  Reasoning and Problem Solving | 0.488 (2.0863) | 1.460 (1.9621)
  Social Cognition | -0.411 (3.0119) | -0.750 (2.7790)
Statistical Analysis 1: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.0225, ANCOVA; Mean Difference (Net) = -4.024, 90% CI 2-sided [-6.872 to -1.175] — For Speed of Processing
Statistical Analysis 2: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.3317, ANCOVA; Mean Difference (Net) = -2.240, 95% CI 2-sided [-6.085 to 1.605] — For Attention/Vigilance
Statistical Analysis 3: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.3243, ANCOVA; Mean Difference (Net) = -2.038, 90% CI 2-sided [-5.482 to 1.406] — For Working Memory
Statistical Analysis 4: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.7497, ANCOVA; Mean Difference (Net) = -0.746, 90% CI 2-sided [-4.667 to 3.175] — For Visual Learning
Statistical Analysis 5: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.1585, ANCOVA; Mean Difference (Net) = 3.112, 90% CI 2-sided [-0.537 to 6.761] — For Verbal Learning
Statistical Analysis 6: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.6582, ANCOVA; Mean Difference (Net) = 0.972, 90% CI 2-sided [-2.709 to 4.654] — For Reasoning and Problem Solving
Statistical Analysis 7: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.9092, ANCOVA; Mean Difference (Net) = -0.338, 90% CI 2-sided [-5.316 to 4.639] — For Social Cognition

5. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale (BPRS) at Week 7
Description: BPRS is the clinician rating of psychiatric symptoms; higher score indicates higher severity; 18-items scored 1-7; lower score is 18 and highest score is 126. The Baseline was calculated as the mean of the second screening assessment and the Day 1 pre-dose assessment. If either measurement meant to be used in the mean was missing, then the Baseline value was the non-missing assessment. If both were missing, then Baseline was considered missing and the task was excluded from the analysis. Change from Baseline was calculated as score at a given time post Baseline minus score at Baseline.
Time Frame: Baseline and Week 7
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 22 | 20
Scores on a scale | -2.795 (1.2410) | -3.819 (1.1512)
Statistical Analysis 1: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.4406, Mixed Model Repeated Measure; Mean Difference (Net) = -1.024, 90% CI 2-sided [-3.237 to 1.190]

6. Secondary Outcome: Change From Baseline in Schedule for Assessment of Negative Symptoms (SANS) at Week 7
Description: The SANS was a tool used to assess five symptom complexes to obtain clinical ratings of negative symptoms in par. with schizophrenia. Complexes include: affective blunting; alogia (impoverished thinking); avolition/apathy; anhedonia/asociality; and disturbance of attention. Assessment was conducted on six-point scale (0=not at all to 5=severe) for a total scoring range of 0-120. Lower scores represent better performance. The Baseline was calculated as the mean of the second screening assessment and the Day 1 pre-dose assessment. If either measurement meant to be used in the mean was missing, then the Baseline value was the non-missing assessment. If both were missing, then Baseline was considered missing and the task was excluded from the analysis. Change from Baseline was calculated as score at a given time post Baseline minus score at Baseline.
Time Frame: Baseline and Week 7
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 22 | 20
Scores on a scale | -3.206 (2.4684) | -5.082 (2.4087)
Statistical Analysis 1: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.5197, Mixed Model Repeated Measure; Mean Difference (Net) = -1.876, 90% CI 2-sided [-6.743 to 2.990]

7. Secondary Outcome: Change From Baseline in University of California and San Diego (UCSD) Performance Based Skills Assessment (UPSA) at Week 7
Description: The UPSA is a measure of Functional Capacity and assesses skills involved in community tasks. It is composed of five subdomains- comprehension and planning, finance, communication, mobility and house management. When combined, measures functional capacity. The comprehension and planning ranges from 0 to 14, the finance ranges from 0 to 11, the communication ranges from 0 to 12, the mobility ranges from 0 to 9, and the house management ranges from 0 to 4. Then a medication management score of 0 to 37 is added. In total, the Assessment is thus scored on a 0 to 87 scale, with higher scores indicating better performance. The Baseline was calculated as the mean of the second screening assessment and the Day 1 pre-dose assessment. If either was missing, then the Baseline value was the non-missing assessment. If both were missing, then Baseline was considered missing and the task was excluded from the analysis. Change from Baseline was score at a given time post Baseline minus Baseline score
Time Frame: Baseline and Week 7
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 22 | 20
Scores on a scale | 2.926 (2.6007) | 4.750 (2.3332)
Statistical Analysis 1: Comparison: Placebo vs GSK239512; Test type: Superiority or Other; p = 0.4637, Mixed Model Repeated Measure; Mean Difference (Net) = 1.824, 90% CI 2-sided [-2.334 to 5.982]

8. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to Day 59
Population: Safety Population consisted of all randomized par. who took at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 25 | 25
Participants
  Any AE | 16 | 17
  Any SAE | 1 | 0

9. Secondary Outcome: Number of Par. With Most Severe On-treatment Abnormal Electrocardiogram (ECG) Findings
Description: Triplicate 12-lead ECGs were obtained at Baseline (screening visit). Single 12-lead ECGs were obtained at each subsequent time point during the study. Abnormal ECG findings were presented for the most severe on-treatment result.
Time Frame: Up to Day 59
Population: Safety Population. Only those participants who showed most severe on-treatment abnormal ECG findings are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 25 | 22
Participants | 8 | 10

10. Secondary Outcome: Number of Par. With Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Readings Outside Clinical Concern Range
Description: Blood pressure readings both systolic and diastolic were collected at pre-dose and then hourly post-dose until 6 hours post-dose or until the par. got discharged. Blood pressure was measured in both standing (Std) and supine (Sup) position. Data with only abnormal values were presented. For SBP the data of concern was <90 or >140 and increase from Baseline (IFB) >=40; <90 or >140 and decrease from Baseline (DFB) >=30. For DBP the data of concern was <50 or >90 and IFB >=30; <50 or >90 and DFB >=20.
Time Frame: Up to Day 59
Population: Safety Population. Only those par. available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 25 | 25
Participants
  SBP, Std, Week 3, <90 or >140 and DFB>=30: number analyzed (Participants) | 23 | 20
  SBP, Std, Week 3, <90 or >140 and DFB>=30 | 1 | 0
  SBP, Std, Week 4, <90 or >140 and DFB>=30: number analyzed (Participants) | 21 | 20
  SBP, Std, Week 4, <90 or >140 and DFB>=30 | 1 | 0
  SBP, Std, Week 5, <90 or >140 and IFB>=40: number analyzed (Participants) | 22 | 20
  SBP, Std, Week 5, <90 or >140 and IFB>=40 | 1 | 0
  SBP, Std, Week 5, <90 or >140 and DFB>=30: number analyzed (Participants) | 22 | 20
  SBP, Std, Week 5, <90 or >140 and DFB>=30 | 1 | 0
  SBP, Std, Week 6, <90 or >140 and DFB>=30: number analyzed (Participants) | 22 | 20
  SBP, Std, Week 6, <90 or >140 and DFB>=30 | 1 | 0
  SBP, Std, follow-up, <90 or >140 and DFB>=30: number analyzed (Participants) | 23 | 24
  SBP, Std, follow-up, <90 or >140 and DFB>=30 | 1 | 0
  SBP, Sup, Week 5, <90 or >140 and IFB>=40: number analyzed (Participants) | 22 | 20
  SBP, Sup, Week 5, <90 or >140 and IFB>=40 | 1 | 0
  DBP, Std, Week 6, <50 or >90 and IBP >=30: number analyzed (Participants) | 22 | 20
  DBP, Std, Week 6, <50 or >90 and IBP >=30 | 1 | 0
  DBP, Sup, Week 6, <50 or >90 and IBP >=30: number analyzed (Participants) | 22 | 20
  DBP, Sup, Week 6, <50 or >90 and IBP >=30 | 1 | 0

11. Secondary Outcome: Number of Par. With Heart Rate Measured Value Outside Clinical Concern Range
Description: Heart rate readings were collected at pre-dose and then hourly post-dose until 6 hours post-dose or until the participant got discharged. It was measured in both supine and standing position. For both Std and Sup positions, heart rate data of concern was <50 or >100 and IFB >=30; <50 or >100 and DFB >=30. Data with only abnormal values were presented.
Time Frame: Up to Day 59
Population: Safety Population. Only those par. available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 25 | 25
Participants
  Std, Week 5, <50 or >100 and IFB >=30: number analyzed (Participants) | 22 | 20
  Std, Week 5, <50 or >100 and IFB >=30 | 1 | 0
  Std, follow-up, <50 or >100 and IFB >=30: number analyzed (Participants) | 23 | 24
  Std, follow-up, <50 or >100 and IFB >=30 | 1 | 0

12. Secondary Outcome: Number of Par. With Abnormal Hematology Parameters Values at Any Time on Treatment
Description: Hematology parameters: Basophils, Eosinophils, Hematocrit, Hemoglobin, Lymphocytes, Mean Corpuscle Hemoglobin (MCH), Mean Corpuscle Hemoglobin concentration (MCHC), Mean Corpuscle Volume (MCV), Monocytes, Platelet count, Red blood cell count (RBC), Reticulocytes, Neutrophils count and White blood cell (WBC) count were presented as values of potential clinical concern at any time on treatment. Only those parameters with any abnormal value are presented.
Time Frame: Up to Day 59
Population: Safety Population. Only those par. available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 25 | 22
Participants
  Eosinophils, Low | 8 | 4
  Eosinophils, High | 1 | 0
  Hemoglobin, Low | 1 | 0
  Monocytes, Low | 3 | 1
  RBC count, Low | 1 | 0
  Reticulocytes, Low | 1 | 1
  Neutrophils count, Low | 1 | 0

13. Secondary Outcome: Number of Par. With Abnormal Clinical Chemistry Parameters Values at Any Time On-treatment
Description: Clinical chemistry parameters: Alanine Amino Transferase (ALT), Albumin, Alkaline Phosphatase, Aspartate Amino Transferase (AST), Calcium, Creatinine, Direct Bilirubin, Gamma Glutamyl Transferase (GGT), Glucose, Potassium, Sodium, Total Bilirubin, Total protein, Urea/ Blood urea nitrogen (BUN) were presented as values of potential clinical concern at any time on treatment. Only those parameters with any abnormal value are presented.
Time Frame: Up to Day 59
Population: Safety Population. Only those par. available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 25 | 22
Participants
  ALT, High | 1 | 3
  AST, High | 1 | 1
  GGT, High | 0 | 3
  Glucose, Low | 2 | 3
  Glucose, High | 5 | 4

14. Secondary Outcome: Number of Par. With Abnormal Urinalysis Parameters Values of Potential Clinical Concern
Description: Samples for urinalysis were collected on Days 1, 7, 14, 21, 28, 35, 42, 49 and up to Day 59 (follow-up) to assess specific gravity, pH, glucose, protein, blood and ketone by dipstick and microscopic examination (if blood or protein is abnormal).
Time Frame: Up to Day 59
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK239512
Number analyzed (Participants) | 25 | 25
Participants | 0 | 0

15. Secondary Outcome: Plasma Concentrations of GSK239512 (Cmax) at Steady State After Repeat Dosing on Dose Review Visit at Any Time On-treatment
Description: One Pharmacokinetic (PK) sample was collected within 15 minutes prior to the start of the CSSB and one PK sample was collected within 15 minutes after completion of the CSSB. 'n' was the number of samples available for analysis.
Time Frame: 15 minutes prior to start and 15 minutes after completion of CSSB at Week 1,2,3,4,5,6 and 7
Population: PK-concentration population included all par. for whom a PK sample was obtained and analyzed. Number of units analyzed are number of samples available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Units Other Than Participants: Plasma sample
Groups:
- GSK239512 10 mcg: Par. received GSK239512 10 mcg daily as dose level 1 in the first week of study.
- GSK239512 20 mcg: Par. received GSK239512 20 mcg daily as dose level 2 in the second week of study.
- GSK239512 40 mcg: Par. received GSK239512 40 mcg daily as dose level 3 in the third week of study.
- GSK239512 80 mcg: Par. received GSK239512 80 mcg daily as dose level 4 in the fourth week of study and continued to receive from fifth to seventh week as maintenance phase.
Arm/Group | GSK239512 10 mcg | GSK239512 20 mcg | GSK239512 40 mcg | GSK239512 80 mcg
Number analyzed (Participants) | 21 | 21 | 21 | 21
Number analyzed (Plasma sample) | 13 | 30 | 11 | 41
nanograms per milliliter (ng/mL) | 0.0250 (37.44) | 0.0496 (29.84) | 0.0790 (51.85) | 0.1775 (42.91)

ADVERSE EVENTS:
Time Frame: All SAEs and non-SAEs were reported up to Day 59.
Description: Safety Population were used to report the AEs and serious AEs.
Groups:
- GSK239512: Par. received oral GSK239512 once daily for a period of 7 weeks (4 weeks titration and 3 weeks at maintenance). Par. started at a daily dose of 10 μg GSK239512 and titrated up weekly through successive dose levels of 20 μg, 40 μg up to a maximum dose of 80 μg according to the titration regimen.
Arm/Group | Placebo | GSK239512
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 11/25 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | GSK239512 (N=25)
Stress (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=25) | GSK239512 (N=25)
Headache (Nervous system disorders) | 4 | 6
Somnolence (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 2
Middle insomnia (Psychiatric disorders) | 2 | 3
Abnormal dreams (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 2
Nightmare (Psychiatric disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.